CLINICAL TRIAL: NCT06186713
Title: Pulmonary Hypertension on Prognosis of Acute Myocardial Infarction Patients With Reduced Left Ventricular Function (STIMULATE): A Single-center, Retrospective Cohort Study
Brief Title: Pulmonary Hypertension on Prognosis of Acute Myocardial Infarction Patients With Reduced Left Ventricular Function
Acronym: STIMULATE
Status: Completed | Type: Observational
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: XJTU1AF2023LSK-406
Record Dates: First submitted 2023-07-06; First posted 2024-01-02 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Acute Myocardial Infarction; Pulmonary Hypertension
Keywords: Acute Myocardial Infarction; Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pulmonary hypertension (PH) group: The PH group comprised of patients with systolic pulmonary artery pressure (sPAP) ≥ 35mmHg measured by echocardiology.
  Interventions: Other: This was an observational study, and no Intervention was given to the patients.
- Control group: The control group included patients with systolic pulmonary artery pressure (sPAP) <35mmHg measured by echocardiology.
  Interventions: Other: This was an observational study, and no Intervention was given to the patients.

INTERVENTIONS:
Other: This was an observational study, and no Intervention was given to the patients. — This was an observational study, and no Intervention was given to the patients.

SUMMARY:
Pulmonary hypertension (PH) has a negative effect on acute myocardial infarction (AMI) patients and appears to be closely associated with reduced left ventricular function. However, its impact on AMI patients with reduced left ventricular function remains unclear. This retrospective study included AMI patients with reduced left ventricular function to investigate the prognostic value of PH in this specific type of patient. Meanwhile, a nomogram would be established basing on the identified independent risk factors, hoping to provide a novel risk stratification for them.

ELIGIBILITY:
Inclusion Criteria:

* The patients who were hospitalized for AMI with reduced left ventricular function at the First Affiliated Hospital of Jiaotong University from January 2018 to January 2022.

Exclusion Criteria:

* Myocardial infarction complicated by cardiac rupture.
* Significant pre-existing heart failure.
* Other comorbidities such as malignancy that may significantly affect prognosis.
* Incomplete clinical data.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This retrospective cohort study included patients who were hospitalized for AMI with reduced left ventricular function at the First Affiliated Hospital of Jiaotong University from January 2018 to January 2022.
Sampling Method: Non-Probability Sample
Enrollment: 4784 (Actual)
Dates: Start 2023-03-30 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
The incidence of all-cause death | 1-year after the AMI.
  All-cause death will be determined by clinical records or phone calls with patients and their family.

CONTACTS AND LOCATIONS:
Overall Officials: Yang Yan, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First Affiliated Hospital of Xian Jiaotong University, Xi'an, Shaanxi, China

REFERENCES:
- [Derived] Liu Q, Zhao C, Dang P, Li Y, Yan Y. Prognostic value of pulmonary hypertension with a nomogram in acute myocardial infarction patients with reduced left ventricular function. Front Cardiovasc Med. 2024 Apr 22;11:1368139. doi: 10.3389/fcvm.2024.1368139. eCollection 2024. PMID 38711791